CLINICAL TRIAL: NCT06795854
Title: Effect of Aerobic Training Versus Relaxation Techniques on Quality of Life in Patients With Post Covid-19 Irritable Bowel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alae Ahmed Salem Ismail, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005264
Record Dates: First submitted 2025-01-26; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Relaxation Therapy; FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic training+ Low fodmap diet (Experimental): This group will include 20 patients. The participants will perform aerobic training (walking on treadmill 25-40 minutes 3 times per week) in addition they will follow a low fodmap diet three times/week for 6 weeks.
  Interventions: Other: Aerobic training; Other: Low fodmap diet
- Relaxation techniques + Low fodmap diet (Experimental): This group will include 20 patients. The participants will perform the relaxation techniques in the form of mindfulness meditation and slow deep breathing in addition they will follow a low fodmap diet for 6 weeks
  Interventions: Other: Relaxation techniques; Other: Low fodmap diet
- Low fodmap diet (Active Comparator): This group will include 20 patients. The participants will receive a low fodmap diet only for 6 weeks.
  Interventions: Other: Low fodmap diet

INTERVENTIONS:
Other: Aerobic training — Sessions will be conducted 3 times per week. Each 40-minute session will include a 5-minute warm-up involving fast walking, slow running, and stretching, followed by an active phase of continuous running. The running period will start at 15 minutes and increase by 2 minutes every two sessions until reaching 30 minutes. The session will conclude with a 5-minute cool-down of slow running and stretching. Exercise intensity will be maintained at 13-15 on the Borg Rate of Perceived Exertion, with continuous walking performed on a treadmill.
  Arms: Aerobic training+ Low fodmap diet
Other: Relaxation techniques — Relaxation techniques will include slow deep breathing and mindfulness meditation exercises. The breathing exercise will involve six cycles per minute, with a 4-second inhalation and a 6-second exhalation, repeated for 30 minutes, three sessions per week. Mindfulness meditation will include a stress and pain management program with sessions starting at 10-15 minutes and gradually increasing to 20-30 minutes, three times per week. Sessions will be conducted in a quiet, comfortable space, focusing on breath awareness, body scanning, thought observation, and optional loving-kindness meditation, concluding with a reflection period.
  Arms: Relaxation techniques + Low fodmap diet
Other: Low fodmap diet — All groups will follow a low-FODMAP diet (LFD). The LFD will exclude foods that commonly aggravate IBS symptoms, such as those containing lactose (dairy), fructose (e.g., apples, pears), and sweeteners like sorbitol and xylitol. Female participants with a BMI of 25 to 29 will aim for a daily calorie intake of 1,800 to 2,200 calories, adjusted based on age, activity level, and metabolism, to maintain weight while managing IBS symptoms effectively.

SUMMARY:
The aim of this study is to compare the effect of aerobic training and relaxation techniques on quality of life in Post covid-19 patients with irritable bowel syndrome .

DETAILED DESCRIPTION:
GI symptoms during active COVID-19 infection increase the chances of developing post-COVID-19 IBS. The risk of developing post-COVID-19 IBS increases in female patients.

The COVID-19 outbreak has caused significant global concern and presents a major challenge for healthcare professionals and public health authorities. Gastrointestinal symptoms are observed in (11-61%) of COVID-19 patients, varying in onset and severity. GI epithelial cells express ACE-2, the primary receptor for SARS-CoV-2.

COVID-19 impacts IBS pathophysiology by disturbing gut microbes. The gut-lung axis, influenced by immune system molecules, often links GI and respiratory disorders.

Post-SARS-CoV-2 infection, IBS prevalence varies by region and study type. In Europe, it's 31%, in North America 16%, and in Asia 7%. A multinational study found a 3% prevalence, cross-sectional studies showed 13%, and longitudinal studies reported 16%.

IBS affects 10-25% of the global population and is a common reason for primary healthcare visits. In the US alone, 2.4-3.5 million people seek medical help yearly for IBS. Recent studies across 38 countries with 395,385 participants reported a 9.2% prevalence. In Western nations, it's 10-18%, while non-Western countries show less attention, with prevalence reaching 35-43% in some developing nations. IBS tends to affect younger individuals more.

IBS is the condition with the highest prevalence among gastrointestinal functional diseases (between 7-10% of the general population, globally).

Prevalence of irritable bowel syndrome by Rome IV. Prevalence of an Internet survey conducted by the Rome Foundation in multiple centers worldwide based on Rome IV. Asia, 1.3%-4.7%; Europe, 3.5%-5.9%; America, 3.5%-5.3%; Australia, 3.5%; Egypt, 7.6%; and South Africa, 5.9%.

IBS prevalence is higher in low- and middle-income countries, particularly among Africans. It increases in the fourth decade by 32.1% and in the fifth decade by 31.1%. Besides known risk factors like female sex, smoking, and stress, previous COVID-19 infection is now recognized as a risk factor. Modifiable risk factors include abnormal BMI, smoking, rich diets, caffeine intake, and low physical activity.

The rising disease rates, particularly in women, require in-depth investigation into their underlying mechanisms. While the exact pathophysiology remains unclear, factors such as altered GI motility, visceral hypersensitivity, microbiota imbalance, brain-gut axis dysfunction, digestive tract inflammation, and psychological factors seem to influence the onset and progression of IBS.

So, the aim of this study is to compare the effect of aerobic training and relaxation techniques on quality of life in Post covid -19 patients with irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index range from 25 to 29.9 kg/m2.
* Patients meeting the Rome IV diagnostic criteria for IBS, it is characterized by the presence of recurrent abdominal pain, on average, at least 1 day a week in the last 3 months with onset of symptoms at least 6 months before diagnosis, associated with 2 or more factors: related to defecation and/or associated with change in stool frequency and/or associated with change in stool form.
* Clinically and medically stable.
* Baseline IBS-SSS score from 75 to 299(mild and moderate).
* No medication for IBS (except for emergencies) within at least 2 weeks ago.
* All patients are not following any type of diet protocol within 3 months prior to the treatment.

Exclusion Criteria:

* The patient has a history of rheumatic diseases in the lower limb.
* Having a history of metabolic, neurologic, cardiovascular, respiratory, renal, and lung problems which would prevent them from participating in aerobic exercises.
* Having a history of knee injury or knee surgery during the past year
* Having a history of fracture in the lower limb during the past six months
* Major vision disorders.
* Hereditary or acquired musculoskeletal disorders in the lower limb.
* Organic gastrointestinal disorders.
* Using drugs that would affect metabolism
* Intestinal organic diseases or systemic diseases affecting gastrointestinal motility (such as gallbladder pancreatitis, hyperthyroidism, diabetes, chronic renal insufficiency, and nervous system diseases).
* History of abdominal or rectal anus surgery.
* Pregnancy or breastfeeding, and post-partum 12 months
* Patient undergoes chemotherapy.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
IBS Severity Scoring System (IBS-SSS) | 6 weeks
  The questionnaire consists of five questions; abdominal pain intensity, abdominal distension, life interference, bowel habit dissatisfaction and abdominal pain frequency. Each item can be scored from 0-100 (according to the value marked by the patient on the visual analog scale or the number of days multiplied by 10), thus the overall IBS severity score ranges from 0 to 500; which according to the original validation can be classified as: < 75 healthy subjects or disease in remission; 75-175 mild disease; 175-300 moderate and > 300 severe disease.
IBS Quality of Life (IBS-QOL) | 6 weeks
  The questionnaire includes 34 question concerning IBS's impact on psychological, social, and daily living activities. The scale can be subdivided into subscales such as dysphoria, activity interference, avoidance of food, health worry, image of body, social, sexual, as well as relationships. Items 1, 2, 4, 8-10, 12, 13, 16, 25-29, and 34 use the following response scale (1=not at all, 2= slightly, 3=moderately, 4=quite a bit, and 5= extremely). Items 3, 5-7, 11, 14, 15, 17-24 and 30- 33 use the following response scale: (1=not at all, 2=slightly, 3=moderately, 4=quite a bit, and 5=a great deal).

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | 6 weeks
  It is used to determine self-reported sleep quality and sleep disturbances for the preceding month. It is a 19-item test and consists of seven components: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) sleep efficiency, (5) sleep disturbance, (6) sleeping medication use and (7) daytime dysfunction. Each component is scored from 0 to 3, and the total score ranges from 0 to 21. The Arabic version of the questionnaire will be used.
Perceived Stress Questionnaire (PSQ) | 6 weeks
  The Perceived Stress Questionnaire (PSQ) assesses an individual's subjective experience of stress, which is crucial for evaluating stress-related symptoms in irritable bowel syndrome (IBS), especially in post-COVID patients. The PSQ includes questions about emotional, time, and social stress, with responses scored on a Likert scale (0-4). Elevated perceived stress is known to exacerbate IBS symptoms, and post-COVID patients often report increased stress due to ongoing health concerns. The PSQ can help identify stress as a key factor in symptom severity, guiding targeted interventions such as stress management techniques (e.g., cognitive behavioral therapy, mindfulness) for better clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Hany Ezzat Obaya, PhD, Study Chair — Assistant Professor, Cairo university
Locations (1):
- Faculty of physical therapy, Cairo University, Giza, Egypt